CLINICAL TRIAL: NCT03177798
Title: Mitochondrial Dysfunction in Chronic Kidney Disease
Brief Title: Mitochondria and Chronic Kidney Disease
Acronym: MitoCKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jorge Gamboa, Research Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 131602
Record Dates: First submitted 2017-05-08; First posted 2017-06-06 (Actual); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Hemodialysis-Induced Symptom; Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases | interventions — icatibant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Icatibant then Placebo (Experimental): Icatibant will be intravenously infused at a rate of 50 ug/kg/h for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours)
  1 week washout
  Placebo will be intravenously infused at the same rate of Icatibant (50 ug/kg/h) for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours)
  Interventions: Drug: Icatibant; Drug: Placebo
- Placebo then Icatibant (Experimental): Placebo will be intravenously infused at the same rate of Icatibant (50 ug/kg/h) for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours)
  1 week washout
  Icatibant will be intravenously infused at a rate of 50 ug/kg/h for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours)
  Interventions: Drug: Icatibant; Drug: Placebo

INTERVENTIONS:
Drug: Icatibant — Subjects will receive either Icatibant or placebo in the first study day. After a washout period of 3 weeks, participant will receive the other treatment. Icatibant (50µg/kg/h) or placebo will be infused for 1 hour prior to the initiation of dialysis and continue through hemodialysis. Hemodialysis session will last approximately 4 hours. Two hours after the end of hemodialysis, The investigators will evaluate mitochondrial function by 31 phosphorus magnetic resonance spectroscopy.
  Other Names: HOE-140
Drug: Placebo — Subjects will receive either Icatibant or placebo in the first study day. After a washout period of 3 weeks, participant will receive the other treatment. Icatibant (50µg/kg/h) or placebo will be infused for 1 hour prior to the initiation of dialysis and continue through hemodialysis. Hemodialysis session will last approximately 4 hours. Two hours after the end of hemodialysis, the investigators will evaluate mitochondrial function by 31 phosphorus magnetic resonance spectroscopy.
  Other Names: placebo infusion

SUMMARY:
The overarching goal of this study is to determine the role of chronic kidney disease and the activation of the kallikrein-kinin system during hemodialysis on the development of mitochondrial dysfunction; the investigators will measure mitochondrial function using the gold standard method, 31-phosphorus magnetic resonance spectroscopy.

The investigators will test the hypothesis that endogenous bradykinin promotes mitochondrial dysfunction in patients undergoing hemodialysis. The investigators will first perform a randomized, placebo-controlled, double-blind, cross-over study measuring the effect of Icatibant (HOE-140), a bradykinin B2 receptor blocker, on mitochondrial function.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have been on maintenance hemodialysis for at least 6 months

Exclusion Criteria:

* History of functional transplant less than 6 months prior to study
* Use of immunosuppressive drugs within 1 month prior to study
* History of active connective tissue disease
* History of acute infectious disease within one month prior to study
* AIDS (HIV seropositivity is not an exclusion criteria)
* History of myocardial infarction or cerebrovascular event within 3 months
* Advanced liver disease
* Gastrointestinal dysfunction requiring parental nutrition
* Active malignancy excluding basal cell carcinoma of the skin
* Ejection fraction less than 30%
* Anticipated live donor kidney transplant
* Pregnancy, breast-feeding or child-bearing potential
* History of poor adherence to hemodialysis or medical regimen
* Subjects with cardiac pacemaker, artificial heart valve, any metallic implant, permanent tattoo, or any retained foreign metallic bodies that are contraindicated in magnetic resonance imaging.
* Inability to provide consent

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cross-over design, eleven individuals receive both treatments, Icatibant and placbo
Groups:
- Icatibant Then Placebo: Icatibant will be intravenously infused at a rate of 50 ug/kg/h for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours).
  Washout, then
  Placebo will be intravenously infused at the same rate of Icatibant (50 ug/kg/h) for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours)
  Two hours after the end of hemodialysis, the investigators will evaluate mitochondrial function by 31 phosphorus magnetic resonance spectroscopy.
- Placebo Then Icatibant: Placebo will be intravenously infused at the same rate of Icatibant (50 ug/kg/h) for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours).
  Washout, then
  Icatibant will be intravenously infused at a rate of 50 ug/kg/h for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours).
  Two hours after the end of hemodialysis, the investigators will evaluate mitochondrial function by 31 phosphorus magnetic resonance spectroscopy.
Period: Overall Study
Arm/Group | Icatibant Then Placebo | Placebo Then Icatibant
Started | 5 | 6
Intervention 1 | 5 | 6
Washout | 5 | 6
Intervention 2 | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients on hemodialysis three times a week for at least six months
Groups:
- Icatibant Then Placebo: Icatibant will be intravenously infused at a rate of 50 ug/kg/h for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours)
  Washout, then
  Placebo will be intravenously infused at the same rate of Icatibant (50 ug/kg/h) for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours)
  Two hours after the end of hemodialysis, the investigators will evaluate mitochondrial function by 31 phosphorus magnetic resonance spectroscopy.
- Placebo Then Icatibant: Placebo will be intravenously infused at the same rate of Icatibant (50 ug/kg/h) for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours).
  Washout, then
  Placebo will be intravenously infused at the same rate of Icatibant (50 ug/kg/h) for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours).
  Two hours after the end of hemodialysis, the investigators will evaluate mitochondrial function by 31 phosphorus magnetic resonance spectroscopy.
- Total: Total of all reporting groups
Arm/Group | Icatibant Then Placebo | Placebo Then Icatibant | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (11.08) | 44.3 (11.32) | 44.73 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 1 | 1 | 2
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Phosphocreatine (PCR) Recovery Time After Knee Extension Assessed by 31 Phosphorus Magnetic Resonance Spectroscopy (31P-MRS)
Description: Mitochondria function will be evaluated using 31P-MRS, which evaluates the concentration of phospho-creatine (PCr) and other phosphate-energy carrier molecules. After basal measurements, subjects will be asked to perform 90 seconds of knee extension followed by 4 minutes of rest. The exercise/rest cycle will be repeated 3 times. Magnetic resonance spectra will be used to calculate concentrations of inorganic phosphate (Pi), PCr, and adenosine triphosphate (ATP). The time constant tau of PCr recovery (time to achieve 66.3% maximal concentration during recovery) will be used to determine mitochondrial function.
Time Frame: Up to 2 hours after completion of drug infusion
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Icatibant: Icatibant will be intravenously infused at a rate of 50 ug/kg/h for 30 minutes prior to the initiation of dialysis and continue through hemodialysis (4 hours)
  Icatibant: Subjects will receive either Icatibant or placebo in the first study day. After a washout period of 3 weeks, participant will receive the other treatment. Icatibant (50µg/kg/h) or placebo will be infused for 1 hour prior to the initiation of dialysis and continue through hemodialysis. Hemodialysis session will last approximately 4 hours. Two hours after the end of hemodialysis, The investigators will evaluate mitochondrial function by 31 phosphorus magnetic resonance spectroscopy.
- Placebo: Placebo will be intravenously infused at the same rate of Icatibant (50 ug/kg/h) for 30 minutes prior to the initiation of dialysis and continue through hemodialysis (4 hours)
  Placebo: Subjects will receive either Icatibant or placebo in the first study day. After a washout period of 3 weeks, participant will receive the other treatment. Icatibant (50µg/kg/h) or placebo will be infused for 1 hour prior to the initiation of dialysis and continue through hemodialysis. Hemodialysis session will last approximately 4 hours. Two hours after the end of hemodialysis, the investigators will evaluate mitochondrial function by 31 phosphorus magnetic resonance spectroscopy.
Arm/Group | Icatibant | Placebo
Number analyzed (Participants) | 11 | 11
seconds | 60.59 (13.94) | 62.66 (29.4)

2. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure will be monitored every 15 minutes, before, during, and after hemodialysis.
Time Frame: 30 minutes before hemodialysis, during dialysis, and up to 1 hour after hemodialysis
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Icatibant: Icatibant will be intravenously infused at a rate of 50 ug/kg/h for 30 minutes prior to the initiation of dialysis and continue through hemodialysis (4 hours). Blood pressure was monitored before, during, and up to 1 hour after the end of the hemodialysis procedure.
- Placebo: Placebo was intravenously infused at the same rate of Icatibant (50 ug/kg/h) for 30 minutes prior to the initiation of dialysis and continue through hemodialysis (4 hours). Blood pressure was monitored before, during, and up to 1 hour after the end of the hemodialysis procedure.
Arm/Group | Icatibant | Placebo
Number analyzed (Participants) | 11 | 11
mmHg
  30 minutes before hemodialysis | 123.36 (15.83) | 125.27 (25.04)
  during dialysis | 122.5454545 (16.87224725) | 122.18 (23.23)
  up to 1 hour after hemodialysis | 119.09 (19.06) | 124.09 (19.90)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Icatibant: Icatibant will be intravenously infused at a rate of 50 ug/kg/h for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours).
  Two hours after the end of hemodialysis, the investigators will evaluate mitochondrial function by 31 phosphorus magnetic resonance spectroscopy.
- Placebo: Placebo will be intravenously infused at the same rate of Icatibant (50 ug/kg/h) for 1 hour prior to the initiation of dialysis and continue through hemodialysis (4 hours).
  Two hours after the end of hemodialysis, the investigators will evaluate mitochondrial function by 31 phosphorus magnetic resonance spectroscopy.
Arm/Group | Icatibant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 2/11
Other Adverse Events (participants affected / at risk) | 1/11 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Icatibant (N=11) | Placebo (N=11)
Hospitalization for cardiac catheterization (Cardiac disorders) | 0 | 1 — Unrelated to the study intervention. Patient require cardiac stent placement due to coronary artery disease
Hypovolemia (Gastrointestinal disorders) | 0 | 1 — Unrelated to the study. Patients was hospitalized due to hypovolemia secondary to gastrointestinal disorders
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icatibant (N=11) | Placebo (N=11)
Patient was admitted for possible kidney transplant (Renal and urinary disorders) | 1 (1) | 0 (0) — Patient did not match and was not eligible for kidney transplant
Arterious venous access thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Unrelated to the the study. Patient had thrombosis of the AV access that requires revascularization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT03177798/Prot_SAP_000.pdf